CLINICAL TRIAL: NCT06430437
Title: A Randomized, Open-Label, Multicenter Phase III Study of SHR-A1811 for First-Line Treatment in Subjects With HER2-Mutated Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of SHR-A1811 in First-line Treatment of Patients With Advanced or Metastatic Non-small Cell Lung Cancer With HER2 Mutations
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-310
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-02

CONDITIONS: Non-Small Cell Lung Cancer With HER2- Mutations
MeSH Terms: interventions — CP protocol; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1811 (Experimental)
  Interventions: Drug: SHR-A1811
- Standard of Care（PD-1/ PD-L1 inhibitors、Pemetrexed/ Paclitaxel、Carboplatin/ Cisplatin） (Active Comparator)
  Interventions: Drug: PD-1/PD-L1 inhibitors、Pemetrexed/ Paclitaxel、Carboplatin/ Cisplatin

INTERVENTIONS:
Drug: SHR-A1811 — Drug: SHR-A1811 administered intravenously every 3 weeks (Q3W)
  Arms: SHR-A1811
Drug: PD-1/PD-L1 inhibitors、Pemetrexed/ Paclitaxel、Carboplatin/ Cisplatin — Drug: PD-1/PD-L1 inhibitors administered intravenously every 3 weeks (Q3W)
  Drug: Pemetrexed Based on the investigator's choice was administered intravenously every 3 weeks (Q3W)
  Drug: Paclitaxel Based on the investigator's choice was administered intravenously every 3 weeks (Q3W)
  Drug: Carboplatin Based on the investigator's choice was administered intravenously every 3 weeks (Q3W)
  Drug: Cisplatin Based on the investigator's choice was administered intravenously every 3 weeks (Q3W)
  Arms: Standard of Care（PD-1/ PD-L1 inhibitors、Pemetrexed/ Paclitaxel、Carboplatin/ Cisplatin）

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of SHR-A1811 versus Standard of Care as first-line treatment of advanced or metastatic Non-Small Cell Lung Cancer with HER2- Mutations

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. 18-75 years old (inclusive of both ends)
3. ECOG score of 0 or 1.
4. Patients with histologically or cytologically confirmed advanced or metastatic NSCLC.
5. Subjects with central laboratory- confirmed functional HER2 mutations
6. No prior systemic antitumor therapy (including investigational agents) for advanced or metastatic NSCLC.
7. Have at least one measurable lesion outside the central nervous system that meets the criteria defined by RECIST v1.1
8. Protocol-defined adequate organ function including cardiac, renal, hepatic function

Exclusion Criteria:

1. Mixed lung cancer with small cell components and sarcomatoid carcinoma confirmed by histology or cytology.
2. Concurrently carrying other driver gene mutations, and targeted drugs for such driver gene mutations have been approved for market release.
3. Subjects with untreated or active metastasis of central nervous system (CNS) tumors, or a history of meningeal metastasis or current meningeal metastasis.
4. With poorly controlled tumor-related pain.
5. previous or current with other malignancies.
6. Subjects with a history of interstitial pneumonia/non-infectious pneumonia requiring hormone therapy, or current interstitial pneumonia/non-infectious pneumonia.
7. Subjects with active or previous autoimmune diseases.
8. Subjects with uncontrolled or severe cardiovascular diseases.
9. Subjects with active hepatitis B or hepatitis C.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) based on blinded independent central review (BICR) | Until progression, assessed up to approximately 2 years
  Defined as time from randomization until progression per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR)

SECONDARY OUTCOMES:
Overall Survival (OS) | Until death, assessed up to approximately 3 years
  Defined as time from randomization until the date of death due to any cause
Progression Free Survival (PFS) by investigator assessment | Until progression, assessed up to approximately 2 years
  Defined as time from randomization until progression per RECIST 1.1 as assessed by the investigator
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) | until to 90 days after the last dose，assessed up to approximately 3 years
  Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided